CLINICAL TRIAL: NCT01802970
Title: Pilot Safety and Blood Immune Cell Transcriptional Profiling Study of Anakinra Plus the Physician's Chemotherapy Choice in Metastatic Breast Cancer Patients
Brief Title: Safety and Blood Immune Cell Study of Anakinra Plus Physician's Chemotherapy Choice in Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 012-099
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Metastatic Breast Cancer
Keywords: Anakinra; Nab Paclitaxel; Capecitabine; Eribulin; Vinorelbin
MeSH Terms: conditions — Breast Neoplasms | interventions — Interleukin 1 Receptor Antagonist Protein; Standard of Care; Capecitabine; eribulin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anakinra plus Standard of Care (Experimental): Patients will undergo a 2-week run-in treatment of daily anakinra alone. This will be followed by daily anakinra (100 mg SC) plus the physician's chemotherapy ( TPC) choice of standard of care (SOC) for a maximum of 6 months.TPC choice includes nab paclitaxel (100 mg/m^2 Intravenous on day 1,8 &15 of a 28 day cycle), or capecitabine (1000mg/m^2 per oral; BID choice: 14 days on, 7 days off OR 7 days on, 7 days off of a 21 day cycle), or eribulin (1.4 mg/m^2 intravenous on day 1 & 8 of a 21 day cycle), or vinorelbine (25mg/m^2 on day 1,8,15 of a 28 day cycle). After 6 months, patients may continue their SOC treatment alone until disease progression or intolerable toxicity.
  Interventions: Drug: Anakinra plus Standard of Care

INTERVENTIONS:
Drug: Anakinra plus Standard of Care — Patients will undergo a 2-week run-in treatment of daily anakinra alone. This will be followed by daily anakinra (100 mg SC) plus the physician's chemotherapy ( TPC) choice of standard of care (SOC) for a maximum of 6 months.TPC choice includes nab paclitaxel (100 mg/m^2 Intravenous on day 1,8 &15 of a 28 day cycle), or capecitabine (1000mg/m^2 per oral; BID choice: 14 days on, 7 days off OR 7 days on, 7 days off of a 21 day cycle), or eribulin (1.4 mg/m^2 intravenous on day 1 & 8 of a 21 day cycle), or vinorelbine (25mg/m^2 on day 1,8,15 of a 28 day cycle). After 6 months, patients may continue their SOC treatment alone until disease progression or intolerable toxicity.
  Other Names: Anakinra: kineret; Nab paclitaxel: Abraxane; Capecitabine: Xeloda; Eribulin: Halaven; Vinorelbine: Navelbine

SUMMARY:
To determine the safety of administering anakinra plus the physician's chemotherapy choice (TPC) of nab paclitaxel, capecitabine, eribulin, or vinorelbine in patients with metastatic breast cancer (MBC), as well as determining blood immune cell transcriptional signatures in patients who undergo IL-1 receptor blockade.

DETAILED DESCRIPTION:
In an attempt to reverse the immune suppressive microenvironment and to enhance chemotherapy effectiveness, decrease tumor metagenicity and decrease IL-1-induced fatigue, metastatic breast cancer (MBC) patients will be treated with chemotherapy plus anakinra. This is a pilot safety, single arm, open label trial. The objective is to determine the safety of anakinra plus the physician's chemotherapy choice (TPC) of nab paclitaxel, capecitabine, eribulin, or vinorelbine in patients with MBC and to define an anakinra-induced anti-IL-1 whole blood transcriptional profile.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients ≥18 years of age.
* Histologically confirmed invasive breast cancer, locally unresectable or metastatic.
* No more than 4 prior chemotherapy regimens for metastatic disease.
* Patients currently being treated with nab paclitaxel, capecitabine,eribulin, or vinorelbine who have had a CR, PR, or SD and who have developed Grade 2, 3, or 4 fatigue on the chemotherapy are eligible for the study. It should be anticipated that these patients will continue to be treated on the same chemotherapy agent for at least 3 more months beyond the time of enrollment.
* Prior hormonal therapy in the adjuvant or metastatic setting is permitted.
* HER2-negative breast cancer. If HER2-, it is defined as follows:

  1. FISH-negative (FISH ratio <2.0), or
  2. IHC 0-1+, or
  3. IHC 2+ AND FISH-negative (FISH ratio<2.0)
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Adequate hematologic function, defined by:

  1. Absolute neutrophil count (ANC) >1500/mm^3
  2. Platelet count ≥100,000/mm^3
  3. Hemoglobin >8 g/dL
* Adequate liver function, defined by:

  1. AST and ALT ≤2.5 x the upper limit of normal (ULN) or ≤5 x ULN in presence of liver metastases
  2. Total bilirubin ≤1.5 x ULN
* Adequate renal function, defined by:

  a. Serum creatinine ≤1.5 x ULN or calculated creatinine clearance of ≥40 ml/min
* Measurable or nonmeasurable disease by RECIST v1.1 criteria
* Life expectancy ≥24 weeks
* Adequate recovery from recent surgery

  1. Major surgical procedure >28 days from study entry
  2. Minor surgical procedure >7 days from study entry (Portacath placement accepted - patients can start treatment <7 days after portacath placement.)
* Patients with previous history of invasive cancers (including breast cancer) are eligible if definitive treatment was completed more than 5 years prior to initiating current study treatment, and there is no evidence of recurrent disease.
* Patient must be accessible for treatment and follow-up.
* All patients must be able to understand the investigational nature of the study and give written informed consent prior to study entry

Exclusion Criteria:

* Patients with active or untreated brain metastases or meningeal metastases are ineligible. Patients who have had brain metastases resected, or have received brain radiation therapy >4 weeks prior to study entry are eligible if they meet all of the following criteria: 1) patient has been off dexamethasone for >2 weeks; 2) no known progression of brain metastasis.
* Previous radiotherapy for metastatic disease completed <2 weeks prior to study treatment initiation.
* Women who are pregnant or lactating. All patients with reproductive potential must agree to use effective contraception from time of study entry until at least 3 months after the last administration of study drug.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation such as: -

  1. severe impaired lung functions as defined as spirometry and DLCO that is 50% of the normal predicted value and/or O2 saturation that is 88% or less at rest on room air
  2. uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN
  3. liver disease such as cirrhosis or severe hepatic impairment (Child-Pugh class C).
* History of any other disease, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug, or that might affect interpretation of the results of this study, or render the subject at high risk for treatment complications.
* Patients may not receive any other investigational treatments while participating in this study.
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Concurrent severe, uncontrolled infection or intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
Safety - Adverse Events in participants | up to 7 months
  Patients will receive anakinra plus the physicians chemotherapy choice of nab paclitaxel, or capecitabine, or eribulin, or vinorelbine for metastatic breast cancer. Adverse events will be recorded throughout the trial, and regardless of the severity will be followed up by investigator until resolution is satisfactory. All adverse events and toxicities will be recorded and assessed for 30 days following the last dose of anakinra at a maximum of 6 months. Grading will be done using Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.

SECONDARY OUTCOMES:
To determine investigator-assessed objective response rate, clinical benefit rate, progression-free survival, and rates of chemotherapy or cancer-related anemia (HgB<10), and an anakinra-induced anti-IL-1 blood transcriptional signatures | upto 7 months
  Objective response rate, clinical benefit rate and progression-free survival in patients will be determined using radiological assessment of tumors (CT/MRI/X-ray/PET), clinical and functional evaluation of patients with 95% confidence intervals. Whole blood transcriptional profiling will be performed to determine a gene expression signature that is induced by IL-1 receptor blockade by anakinra. The gene expression signatures from baseline will be compared to those signatures obtained after the 2-week run-in treatment with anakinra alone. During the treatment, complete blood count with differential/platelet count and complete metabolic profiling will be done to identify any baseline changes.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce O'Shaughnessy, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States